CLINICAL TRIAL: NCT03891225
Title: Efficacy of Amniotic Membrane Implantation Over Pancreo-jejunal Anastomosis After Pancreaticoduodenectomy in Reducing Post-operative Pancreatic Fistula POPF.
Brief Title: Efficacy of Amniotic Membrane Over Pancreatic Anastomosis After Pancreaticoduodenenctomy to Preventing Pancreatic Fistula
Acronym: POPF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Casa di Cura Dott. Pederzoli (Other)
Collaborators: Fondazione Banca dei Tessuti di Treviso onlus (Unknown)
Responsible Party: Principal Investigator, Isabella Frigerio, MD, PhD, Principal Investigator, Casa di Cura Dott. Pederzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2039CESC
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Post Operative Pancreatic Fistula; Pancreatic Resection; Biological Dressing

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amniotic Membrane implantation Arm (Experimental): All consecutive patients undergone pancreaticoduodenectomy with high FRS will be treated with implantation of AM, by overlapping it over the pancreo-jejunal anastomosis.
  Interventions: Procedure: Amniotic Membrane implantation

INTERVENTIONS:
Procedure: Amniotic Membrane implantation — Surgical procedure will be performed with Longemire Traverso technique. At the end of all pancreatic, biliary and duodenal anastomosis, the AM will be implanted.

SUMMARY:
Post-operative pancreatic fistula (POPF) after pancreatic resection is a potentially life-threatening complication occuring in up to 27% of patients undergoing a pancreatic resection. Despite several strategies have been proposed further improvements are needed. Many studies suggest that amniotic membrane(AM) implantation is effective in tissue regeneration and prevention of fluid leakage at many surgical sites. However,the implantation of AM has never been used in pancreatic surgery.

After having completed the first case of implantation of AM we proceed with this pilot study to determine in 20 consecutive patients undergone to pancreaticoduodenectomy (PD) with high risk of POPF, the efficacy of AM in reducing this event and the related morbidity.

DETAILED DESCRIPTION:
Twenty consecutive patients candidated to PD regardless the diagnosis will be enrolled if presenting an high Fistula Risk Score. Enrollement will be done in O.R. after frozen section of the pancreas. The AM is provided by Fondazione Banca dei Tessuti di Treviso Onlus. The placenta is sourced from donors undergoing caesarean sections and processed shortly after retrieval, donors are evaluated according to Italian requirements. The AM is carefully detached from the chorion and rinsed with sterile saline solution, flattened on a nitrocellulose membrane filter (Merck Millipore), with its stromal side facing down, in contact with the filter. The AM is then immersed in a cocktail of antibiotics then cut into patches and immersed in cryopreservant solution. Cryopreservation was achieved using a programmable cryogenic freezer (Planer KryoSave Integra, 750-30), which triggers a controlled cooling rate. The AM patches were stored in vapor-phase liquid nitrogen. Thirty minutes before its use, the AM was defrozen and washed with saline. A 10x15cm MA patch was placed around the pancreatic anastomoses starting from the posterior surface. The caudal and the cranial flap were overlapped on the anterior surface to wrap the anastomosis. The membrane was than fixed with 4-0 Monocryl sutures at the jejunal surface and at the peri-pancreatic tissue. Then an end-to-side bilio-enteric anastomosis was carried out. The reconstruction was completed by an end-to-side antecolic duodenojejunostomy. At the end of the procedure, two drains were placed ventral and dorsal to the PJ, without friction with the AM.

In the postoperative period will be evaluated: morbidity according to Clavien Dindo classification with attention to clinical relevant pancreatic fistula, bleeding, need of reintervention, surgical site infection, multi drug resistant infection and mortality. Costs and postoperative staying will be monitored as well.

Student t test, Mann Whitney and Chi square will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Undergone to Pancreatico-duodenectomy with high FRS (>=5)
* Adeguate consent

Exclusion Criteria:

* Total pancreatectomy
* Pancreatic anastomosis different from pancreo-jejunal anastomosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
postoperative complications | up to 90 days after surgery
  clinical relevant pancreatic fistula, intra-abdominal collection, acute pancreatitis, SSI, need for reintervention, mortality

SECONDARY OUTCOMES:
correlation between microscopic pancreatic fibrosis and CR POPF | 90 days from surgery
  the absence of microscopic fibrosis in a macroscopically soft pancreas may be related to higher risk of CR POPF and therefore may suggest implementation of anastomotic protecion (ie. the AM)

CONTACTS AND LOCATIONS:
Overall Officials: ISABELLA FRIGERIO, Principal Investigator — PEDERZOLI HOSPITAL
Locations (1):
- Pederzoli Hospital, Peschiera del Garda, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided
UPON REQUEST

REFERENCES:
- [Background] Pulvirenti A, Marchegiani G, Pea A, Allegrini V, Esposito A, Casetti L, Landoni L, Malleo G, Salvia R, Bassi C. Clinical Implications of the 2016 International Study Group on Pancreatic Surgery Definition and Grading of Postoperative Pancreatic Fistula on 775 Consecutive Pancreatic Resections. Ann Surg. 2018 Dec;268(6):1069-1075. doi: 10.1097/SLA.0000000000002362. PMID 28678062
- [Background] McMillan MT, Vollmer CM Jr, Asbun HJ, Ball CG, Bassi C, Beane JD, Berger AC, Bloomston M, Callery MP, Christein JD, Dixon E, Drebin JA, Castillo CF, Fisher WE, Fong ZV, Haverick E, House MG, Hughes SJ, Kent TS, Kunstman JW, Malleo G, McElhany AL, Salem RR, Soares K, Sprys MH, Valero V 3rd, Watkins AA, Wolfgang CL, Behrman SW. The Characterization and Prediction of ISGPF Grade C Fistulas Following Pancreatoduodenectomy. J Gastrointest Surg. 2016 Feb;20(2):262-76. doi: 10.1007/s11605-015-2884-2. Epub 2015 Jul 11. PMID 26162925
- [Background] Patel K, Teta A, Sukharamwala P, Thoens J, Szuchmacher M, DeVito P. External pancreatic duct stent reduces pancreatic fistula: a meta-analysis and systematic review. Int J Surg. 2014;12(8):827-32. doi: 10.1016/j.ijsu.2014.06.008. Epub 2014 Jul 6. PMID 25003575
- [Background] Callery MP, Pratt WB, Kent TS, Chaikof EL, Vollmer CM Jr. A prospectively validated clinical risk score accurately predicts pancreatic fistula after pancreatoduodenectomy. J Am Coll Surg. 2013 Jan;216(1):1-14. doi: 10.1016/j.jamcollsurg.2012.09.002. Epub 2012 Nov 2. PMID 23122535
- [Background] Lin SD, Lai CS, Hou MF, Yang CC. Amnion overlay meshed skin autograft. Burns Incl Therm Inj. 1985 Jun;11(5):374-8. doi: 10.1016/0305-4179(85)90102-0. PMID 3896420
- [Background] Talmi YP, Sigler L, Inge E, Finkelstein Y, Zohar Y. Antibacterial properties of human amniotic membranes. Placenta. 1991 May-Jun;12(3):285-8. doi: 10.1016/0143-4004(91)90010-d. PMID 1754577
- [Background] Barski D, Gerullis H, Ecke T, Varga G, Boros M, Pintelon I, Timmermans JP, Winter A, Bagner JW, Otto T. Repair of a vesico-vaginal fistula with amniotic membrane - Step 1 of the IDEAL recommendations of surgical innovation. Cent European J Urol. 2015;68(4):459-61. doi: 10.5173/ceju.2015.683. Epub 2015 Nov 13. PMID 26855802
- [Background] Knight BC, Kausar A, Manu M, Ammori BA, Sherlock DJ, O'Reilly DA. Evaluation of surgical outcome scores according to ISGPS definitions in patients undergoing pancreatic resection. Dig Surg. 2010;27(5):367-74. doi: 10.1159/000313693. Epub 2010 Oct 13. PMID 20938180